CLINICAL TRIAL: NCT06082791
Title: A Clinical Validation Study to Evaluate the Diagnostic Accuracy of a Cough-based Auxiliary Diagnosis Algorithm for Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Clinical Validation Study to Evaluate the Diagnostic Accuracy of a Cough-based Auxiliary Diagnosis Algorithm for COPD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-199
Record Dates: First submitted 2023-10-08; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-09

CONDITIONS: COPD; Cough; Algorithm
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COPD
- other respiratory disease without COPD
- healthy people without respiratory disease

SUMMARY:
Cough is one of the most common symptoms in COPD patients, and its different characteristics in amplitude, frequency and waveform can be analyzed by intelligent algorithms for the auxiliary diagnosis of COPD. The current study is to conduct external clinical validation of COPD auxiliary diagnosis algorithm and lung function prediction algorithm, and preliminatively verify the performance of the algorithm, with the ultimate goal of developing a portable and rapid COPD auxiliary diagnosis and condition assessment tool that can be used at home.

ELIGIBILITY:
Inclusion Criteria:

* patients with stable COPD were recruited for this study. Inclusion criteria were age ≥40 years and a diagnosis of COPD

Exclusion Criteria:

* Exclusion criteria were acute exacerbations of respiratory symptoms within the past 2 weeks or significant comorbid cardiovascular, neurological, musculoskeletal, immunological, or infectious diseases.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: three cohorts are included COPD respiratory disease without cold healthy people
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Positive Agreement Rate (PPA) | 12.30.2024
  Positive Agreement Rate (PPA) of auxiliary Diagnosis Algorithm for COPD

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes